CLINICAL TRIAL: NCT00536159
Title: Improving the Health and Development of Low-Income Pregnant Women
Brief Title: Medicaid Enhanced Prenatal/Postnatal Services Using a Nurse-Community Health Worker Team
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Corewell Health West (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R50 MC00045-04 R2
Record Dates: First submitted 2007-09-18; First posted 2007-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Perinatal Depression; Stress; Prenatal Health Risk Behaviors; Child Development
Keywords: nurse-community health worker team; perinatal depression; stress; Medicaid enhanced prenatal programs

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Care (Active Comparator): Medicaid eligible/insured pregnant women and their infants are eligible for risk assessment and up to 18 home visits (9/pregnancy and 9/infancy) from community professional providers as part of a state-sponsored enhanced prenatal and postnatal Medicaid program.
  Interventions: Other: Medicaid Maternal and Infant Support Services
- Nurse-CHW Team (Experimental): Nurse-CHW team provided both nursing care, with additional focus on mental health and stress, and intensive relationship-based support from a CHW similar in characteristics to women served in the context of state-sponsored Medicaid program.
  Interventions: Other: Nurse-CHW team

INTERVENTIONS:
Other: Medicaid Maternal and Infant Support Services — Enhanced services include home visiting, transportation, psychosocial counseling, multidisciplinary planning, case management, nutritional guidance, and pregnancy and parenting education during pregnancy and infancy. The services are delivered primarily by nurses with occasional visits by social workers or nutritionists. In the county of the study (Kent), women who were assessed were provided intervention services.
  Arms: Community Care
Other: Nurse-CHW team — A nurse and two CHWs functioned as a team, using visit and clinical guidelines that detailed expected care. Each team provided services for approximately 50-60 families. While occasional visits were made by both providers, most visits were made by either provider alone. Nurses guided the CHW care, led a multidisciplinary team assessment (with social workers, nutritionists, and others), provided crisis intervention and case management, assessed and managed health problems (including screening for depression and mental health care), and had periodic office visits with prenatal providers. CHWs provided relationship-based support by attempting weekly prenatal contact that alternated phone and face-to-face visits and used peer role modeling and personal empowerment approaches.
  Arms: Nurse-CHW Team

SUMMARY:
Our objective was to test whether there were advantages to Nurse-CHW team home visiting designed to combine the strengths of both visitors, with a focus on maternal stress and mental health, when compared with standard of Community Care (CC) that included professional home visitors in a state-sponsored Medicaid program. We conducted the study under usual community conditions in a population of women eligible for state-sponsored Medicaid programs. We predicted that during pregnancy and infancy, women in the Nurse-CHW team intervention would report 1) less perceived stress; 2) fewer depressive symptoms; and 3) increased levels of psychosocial resources (self-esteem, mastery, and social support) than women in CC. Benefits were expected to be most pronounced for women with low psychosocial resources and high stress at enrollment.

DETAILED DESCRIPTION:
Impoverished pregnant and parenting women have greater exposure to environmental stress with adverse effects for their own mental and physical health that may have long term consequences for their children's health and development. The mental health consequences of stress are pervasive in low income pregnant women and mothers with almost half screening positive for depressive symptoms and a quarter meeting diagnostic criteria for major or minor depression. While national home visiting models have demonstrated improvement in health, developmental, and parenting outcomes for women willing to participate, they have had less success in reducing depressive symptoms during pre and postnatal periods, and often programs struggle to engage women with unmet mental health needs.

We conducted a community-based, multi-site, randomized, controlled trial that included longitudinal assessment on five occasions during pregnancy and infancy to determine temporal program effects. We used a CC comparison group because Medicaid insured women in Michigan are eligible for home visiting through enhanced prenatal and infant services, and our goal was to determine if there was any advantage to the team approach when compared to community implementation of the state-sponsored home visiting program.

Pregnant women, who telephoned one of five public clinics in Kent County, Michigan, a county that includes urban (Grand Rapids) and rural areas, were contacted and invited to participate in the trial. We enrolled women considered harder to reach with cultural, language, and literacy barriers to participation and with chronic or current medical problems-populations traditionally served by state-sponsored programs. Participation was not dependent on women coming to a research or health facility, participating in prenatal or child health care or the enhanced services, having reliable transportation, consistent phone service, or stable housing.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid eligible
* residency in the county and no plans to move within 18 months
* at least 16 years of age
* speaks Spanish or English

Exclusion Criteria:

* no pre-existing relationship with a home visiting nurse
* no diagnosis or treatment for a pre-existing mental health condition within the last two years

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 1997-01; Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
depressive symptoms | <24 weeks gestation to 12 months post birth
perceived stress | <24 weeks gestation to 12 months post birth
mastery | <24 weeks gestation to 12 months postbirth
self esteem | <24 weeks gestation to 12 months post birth
social support | <24 weeks gestation to 12 months postbirth

SECONDARY OUTCOMES:
infant motor, mental development | 6 and 12 months postbirth
maternal-infant interaction | 6 and 12 months postbirth
Medicaid (maternal and infant)and program costs | <24 weeks gestation to 12 months
health risk behaviors (smoking, drug, alcohol) | <24 weeks gestation to 12 months postbirth

CONTACTS AND LOCATIONS:
Overall Officials: Lee Anne Roman, MSN, PhD, Principal Investigator — Michigan State University
Locations (1):
- Spectrum Health Hospitals, Grand Rapids, Michigan, United States

REFERENCES:
- [Background] Roman LA, Lindsay JK, Moore JS, Duthie PA, Peck C, Barton LR, Gebben MR, Baer LJ. Addressing mental health and stress in Medicaid-insured pregnant women using a nurse-community health worker home visiting team. Public Health Nurs. 2007 May-Jun;24(3):239-48. doi: 10.1111/j.1525-1446.2007.00630.x. PMID 17456125